CLINICAL TRIAL: NCT01681563
Title: A Single-arm Multi-center Trial of Pentostatin Plus Cyclophosphamide With Ofatumumab (PCO) in Older Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Trial of Pentostatin Plus Cyclophosphamide With Ofatumumab (PCO) in Older Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Collaborators: Regione Lombardia (Other); GlaxoSmithKline (Industry); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCO; 2010-022332-37 (EudraCT Number)
Record Dates: First submitted 2012-06-18; First posted 2012-09-10 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Pentostatin; Cyclophosphamide; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pentostatin/Cyclophosphamide/Ofatumumab (Experimental): Subjects will receive up to 6 cycles of pentostatin, cyclophosphamide, and ofatumumab given every 21 days (+/- 4 days).
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Drug: Ofatumumab

INTERVENTIONS:
Drug: Pentostatin — Lyophilized powder for intravenous administration.
  Other Names: Nipent 10 mg
Drug: Cyclophosphamide — IV
Drug: Ofatumumab — Liquid concentrate for solution for infusion.
  Other Names: Arzerra 100 mg

SUMMARY:
This is a phase II multicenter, non-comparative, open label study in older previously untreated Chronic Lymphocytic Leukaemia patients, requiring therapy, aimed at defining the efficacy profile (ORR, CRR and TTP) of pentostatin and cyclophosphamide given in combination with Ofatumumab (PCO).

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common of the chronic lymphoid leukemias, comprising 30% of all adult leukemias. The majority of CLL patients are of advanced age. Currently, immunochemotherapy with Rituximab, Fludarabine and Cyclophosphamide (RFC) is the standard of care in previously untreated patients with CLL requiring treatment. The combination of Pentostatin and Cyclophosphamide has generated excellent clinical response rates in pretreated B-CLL patients. Early data on the use of Ofatumumab as a single agent in Fludarabine-refractory CLL patients have been reported. Given the reported efficacy of chemo-immunotherapy combinations in CLL and the promising activity and toxicity profile of Pentostatin combinations, we designed a trial of Pentostatin, Cyclophosphamide, and Ofatumumab for previously untreated older patients with CLL. The aim is improving efficacy, in Rituximab resistant CLL, and toxicity considering the good profile of tolerability showed using Ofatumumab as single agent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-CLL defined by:

  1. Circulating lymphocytes of more than or equal to 5 x109/L B lymphocytes (5000/mL) in the peripheral blood for the duration of at least 3 months. AND
  2. Flow cytometry confirmation of immunophenotype: CD5, CD19, CD20, CD23, CD79b, and surface Ig
* Age ≥ 65 years
* Active disease and indication for treatment based on modified NCI-WG guidelines defined by presenting at least any one of the following conditions:
* Evidence of progressive marrow failure as manifested by development of, or worsening of anemia and/or thrombocytopenia
* Massive (i.e. > 6 cm below the left costal margin) or progressive or symptomatic splenomegaly
* Massive nodes (i.e. > 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy
* Progressive lymphocytosis with an increase of > 50% over a two month period or an lymphocyte doubling time < 6 months
* A minimum of any one of the following disease-related symptoms must be present:

  1. Unintentional Weight loss ³ 10% within the previous six months
  2. Fevers > 38.0 °C for ≥ 2 weeks without evidence of infection
  3. Night sweats for more than 1 month without evidence of infection
* Not been previously treated for B-CLL (prior autoimmune hemolytic anemia treatment permitted)
* ECOG Performance Status of 0-2
* Signed written informed consent prior to performing any study-specific procedures

Exclusion Criteria:

* Prior therapy for B-CLL with any agent except corticosteroids used to treat autoimmune hemolytic anemia
* Active autoimmune hemolytic anemia (AIHA) requiring corticosteroid therapy > 100 mg equivalent to hydrocortisone, or chemotherapy
* Known Richter transformation
* Known CNS involvement of B-CLL
* Any radiation therapy ≤ 4 weeks prior to registration;
* Any major surgery ≤ 4 weeks prior to registration;
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C
* Past or current malignancy with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix or the breast unless the tumor was successfully treated with curative intend at least 2 years prior to trial entry.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to Visit 1, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities
* History of significant cerebrovascular disease
* Glucocorticoid unless given in doses ≤ 100 mg/day hydrocortisone (or equivalent dose of other glucocorticoid) if for exacerbations other than B-CLL (e.g. asthma)
* Known HIV positive
* Positive serology for Hepatitis B (HB), defined as a positive test for HBsAg. In addition if negative for HBsAg but HBcAb positive and HBsAb negative a HB DNA test will be performed and if positive the subject will be excluded. Note: if HBcAb positive and HBsAb positive, which is indicative of a past infection, the subject can be included.
* Screening laboratory values:

  1. Creatinine Clearance < 60 mL/min
  2. Total bilirubin > 2.0 times upper normal limit (unless due to liver involvement of BCLL)
  3. ALT > 3.0 times upper normal limit (unless due to liver involvement of B-CLL)
* Treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to Visit 1 or currently participating in any other interventional clinical study
* Known or suspected inability to comply with the study protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 2 months after the last dose received (End of treatment period)
  To assess the overall response rate (ORR) using pentostatin, cyclophosphamide, and ofatumumab in patients with previously untreated CLL requiring therapy.

SECONDARY OUTCOMES:
Adverse Events according to CTCAE, Version 3.0 NCI CTCAE | From informed consent signed through to 28 days after the last study drug administration
  To monitor and assess toxicity of pentostatin, cyclophosphamide, and ofatumumab in patients with previously untreated CLL.
Complete Response Rate (CRR) | Baseline, at cycle 3 and 2 months after the last dose received
  To assess the complete response of CLL patients treated with pentostatin, cyclophosphamide, and ofatumumab
Minimal Residual Disease (MRD) | Every 3 months from the last dose of treatment up to 2 years follow up.
  To determine the proportion of patients who achieve a minimal residual disease (MRD) negative state as assessed by flow cytometry.It will be assessed only in patients responding to PCO treatment.
Progression-Free Survival | Measured as the time from inclusion in the trial to disease progression or death, assessed up to 2 years
  To determine the progression-free survival in CLL patients treated with pentostatin,cyclophosphamide, and ofatumumab.
Overall Survival (OS) | Measured as the time from inclusion in the trial until death from any cause, assessed up to 2 years of follow up
  To assess overall survival (OS) of CLL patients treated with pentostatin, cyclophosphamide, and ofatumumab
Time To Progression (TTP) | Measured as the time from inclusion in the trial until disease progression or death, assessed up to 2 years
  To assess the time-to-progression (TTP) of CLL patients treated with pentostatin, cyclophosphamide, and ofatumumab
Genetic analysis by Fish | Baseline, 2 months after the last dose received and at month 12 and 24 during follow up
  To determine if cytogenetic abnormalities identified by FISH, relate to response to PCO therapy.
Ofatumumab pharmacokinetics parameter | Cycle1: Day 1, 2, 3, 8, 9, 15. Cycles 2-5: Day 1, 2, 3, 8,15. Cycle 6: Day 1, 2, 3, 8, 15, 21
  To assess ofatumumab pharmacokinetic parameters
IgVH mutation status | Baseline, 2 months after the last dose received and at month 12 and 24 during follow up
  To determine if IgVH mutation status relate to response to PCO therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montillo, MD, Study Director — Ospedale Cà Granda - Niguarda S.C: Ematologia; Agostino Cortelezzi, MD, Principal Investigator — Ospedale Maggiore Policlinico Università di Milano Istituto di Ematologia; Giovanni Ucci, MD, Principal Investigator — ASL della provincia di Lodi Presidio Ospedaliero di Lodi Dipartimento di Medicina Interna; Ester Orlandi, MD, Principal Investigator — IRCCS Policlinico San Matteo Pavia Istituto di Ematologia; Fausto Rossini, MD, Principal Investigator — Azienda Ospedaliera San Gerardo di Monza U.O. Ematologia; Armando Santoro, MD, Principal Investigator — IRCCS Istituto Clinico Humanitas di Rozzano Dipartimento di Ematologia; Paolo Ghia, MD, Principal Investigator — IRCCS Ospedale S. Raffaele Università Vita-Salute Dipartimento di Medicina Interna; Marina Motta, MD, Principal Investigator — Presidi Ospedalieri Spedali Civili di Brescia Divisione di Ematologia; Gianluca Gaidano, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Maggiore della Carità - Struttura Complessa a Direzione Universitaria (SCDU Ematologia); Mauro Turrini, MD, Principal Investigator — Ospedale Valduce S.C. Medicina Interna Sezione di Ematologia; Pierangelo Spedini, MD, Principal Investigator — Istituti Ospitalieri di Cremona U.O.Complessa di Ematologia e CTMO; Marta Coscia, MD, Principal Investigator — AOU Città della Salute e della Scienza Ospedale Molinette Divisione di Ematologia; Antonino Mazzone, MD, Principal Investigator — Azienda Ospedaliera Ospedale Civile di Legnano U.O. Medicina Interna; Alessandro Rambaldi, MD, Principal Investigator — A.O. Papa Giovanni XXIII di Bergamo USC Ematologia
Locations (12):
- Italy (12):
  - Azienda Ospedaliera San Gerardo di Monza U.O. Ematologia, Monza, MB
  - IRCCS Istituto clinico Humanitas di Rozzano Dipartimento di Ematologia, Rozzano, Milano
  - Azienda Ospedaliera Ospedale Civile di Legnano U.O. Medicina Interna, Legnano, MI
  - A.O. Papa Giovanni XXIII U.S.C. Ematologia, Bergamo
  - Presidi Ospedalieri Spedali Civili di Brescia Divisione di Ematologia, Brescia
  - Ospedale Valduce S.C. Medicina Interna Sez. Ematologia, Como
  - Ospedale Maggiore Policlinico Università di Milano Istituto di Ematologia, Milan
  - IRCCS Fondazione Centro S. Raffaele del Monte Tabor Università Vita-Salute Dipartimento di Medicina Interna, Milan
  - Ospedale Cà Granda - Niguarda S.C: Ematologia, Milan
  - Azienda ospedaliera-universitaria Maggiore della Carità SCDU Ematologia, Novara
  - IRCCS Policlinico San Matteo Pavia Istituto di Ematologia, Pavia
  - A.O.U. Città della Salute e della Scienza Ospedale Molinette Divisione di Ematologia, Torino

REFERENCES:
- [Derived] Tedeschi A, Rossi D, Motta M, Quaresmini G, Rossi M, Coscia M, Anastasia A, Rossini F, Cortelezzi A, Nador G, Scarfo L, Cairoli R, Frustaci AM, Dalceggio D, Picardi P, De Paoli L, Orlandi E, Rambaldi A, Massaia M, Gaidano G, Montillo M; Rete Ematologica Lombarda-CLL Workgroup. A phase II multi-center trial of pentostatin plus cyclophosphamide with ofatumumab in older previously untreated chronic lymphocytic leukemia patients. Haematologica. 2015 Dec;100(12):e501-4. doi: 10.3324/haematol.2015.132035. Epub 2015 Aug 20. No abstract available. PMID 26294723